CLINICAL TRIAL: NCT02591433
Title: Pilot Study of the Effectiveness of the JeffQuit Smoking Cessation Program
Brief Title: JeffQuit Group Therapy Program for Smoking Cessation in Patients With a History of Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 13D.423; JT 2686 (Other: JeffTrial Number)
Record Dates: First submitted 2015-10-28; First posted 2015-10-29 (Estimated); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Current Smoker; Malignant Neoplasm
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Supportive care (JeffQuit group therapy) (Experimental): Patients undergo three, 1-hour group therapy sessions held by a JeffQuit practitioner over a 1-month period. Patients receive strategies for managing the psychological, habitual, and physiological components of smoking and help with developing a planned quit date. Patients are also provided with advice on how to switch to cigarette brands with less nicotine and then how to substitute the nicotine patch and gum for cigarettes. The JeffQuit counselor is available for additional individual support as needed.
  Interventions: Other: Tobacco Cessation Counseling; Other: Support Group Therapy; Other: Quality-of-Life Assessment

INTERVENTIONS:
Other: Tobacco Cessation Counseling — Undergo JeffQuit group therapy
  Other Names: Tobacco Cessation Counseling, Tobacco Counseling
Other: Support Group Therapy — Undergo JeffQuit group therapy
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment, Quality-of-Life Assessment

SUMMARY:
This pilot clinical trial studies how well the "JeffQuit" group therapy program works in enabling patients with a history of cancer to quit smoking. The JeffQuit program uses group therapy to provide psychological support and address the mental need for smoking, the habit or routine it creates, and the physical need for nicotine. It is not yet known how well the JeffQuit program will work in helping patients with a history of cancer to stop smoking.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the initial effectiveness of the JeffQuit program on smoking cessation in cancer patients.

II. To assess the quality of life improvements related to the JeffQuit smoking cessation program in cancer patients.

OUTLINE:

Patients undergo three, 1-hour group therapy sessions held by a JeffQuit practitioner over a 1-month period. Patients receive strategies for managing the psychological, habitual, and physiological components of smoking and help with developing a planned quit date. Patients are also provided with advice on how to switch to cigarette brands with less nicotine and then how to substitute the nicotine patch and gum for cigarettes. The JeffQuit counselor is available for additional individual support as needed.

After completion of study, patients are followed up at 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. History of cancer
2. Current smoker
3. Willing to provide consent and participate in the JeffQuit program
4. Referral by a Kimmel Cancer Center provider

Exclusion Criteria:

1. Any significant active medical disorder or physical condition that could reasonably be expected to interfere with the ability of the patient to quit smoking as determined by the Principal Investigator (PI)
2. Currently participating in another smoking cessation program
3. Currently receiving chemotherapy or radiation therapy that would interfere with their ability to participate in the JeffQuit program
4. Patients with evidence of a significant psychiatric disorder by history/examination that would prevent completion of the study will not be allowed to participate
5. Patients with current alcohol or drug abuse
6. Enrollment in active clinical trial/ experimental therapy within the prior 30 days
7. Are in the terminal stages of illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-08; Primary Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who are adherent to smoking abstinence | Up to 6 months after completion of intervention
  Calculated along with a 1-sided 95% exact confidence interval. An exact binomial test (with a one-sided alpha of 0.05) will also be used to test whether adherence is greater than 60%.

SECONDARY OUTCOMES:
Change in Patient Reported Outcomes Measurement Information System (PROMIS) quality of life scores | Baseline to up to 6 months after completion of intervention
  The scores for the Patient Reported Outcomes Measurement Information System (PROMIS) questionnaire will be evaluated for differences between the pre and post program states using analysis of variance using mixed models to allow for inclusion of all subjects with at least one measurement, with assessment of post-treatment to pre-treatment changes as the primary consideration. Longitudinal repeated measures using linear mixed models will be applied to assess the change from baseline as the outcome, and an exploratory analysis of potential clinical and demographic modifiers will be completed.
Change in Smoking Cessation Quality of Life (SCQoL) questionnaire scores | Baseline to up to 6 months after completion of intervention
  The scores for the Smoking Cessation Quality of Life (SCQoL) questionnaire will be evaluated for differences between the pre and post program states using analysis of variance using mixed models to allow for inclusion of all subjects with at least one measurement, with assessment of post-treatment to pre-treatment changes as the primary consideration. Longitudinal repeated measures using linear mixed models will be applied to assess the change from baseline as the outcome, and an exploratory analysis of potential clinical and demographic modifiers will be completed.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Newberg, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Sidney Kimmel Cancer Center at Thomas Jefferson University, an NCI-Designated Cancer Center — http://kimmelcancercenter.org
- See also: Jefferson University Hospitals — http://hospitals.jefferson.edu/